CLINICAL TRIAL: NCT03579004
Title: Neoadjuvant Chemotherapy Followed by Preoperative Chemoradiation in Resectable Squamous-cell Esophageal Cancer: Single Arm Phase II Study
Brief Title: Neoadjuvant Chemotherapy Followed by Preoperative Chemoradiation in Resectable Squamous-cell Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mona Frolova (Other)
Responsible Party: Sponsor-Investigator, Mona Frolova, Senior Staff Member, Russian Academy of Medical Sciences
Organization: Russian Academy of Medical Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-038
Record Dates: First submitted 2018-06-12; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Esophageal Neoplasms; Squamous Cell Carcinoma; Concurrent Chemoradiotherapy
Keywords: esophageal squamous cell carcinoma; preoperative chemoradiotherapy; preoperative chemotherapy
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Drug Therapy; Cisplatin; Fluorouracil; Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trimodality approach (Experimental): 2 cycles of neoadjuvant chemotherapy (paclitaxel 175 mg/м2 iv day 1, cisplatin 75 mg/м2 iv day 1, fluorouracil 750 mg/m2/day continuous infusion, day 1-4 every 3 weeks). 3-4 weeks later - preoperative chemoradiotherapy (paclitaxel 50 mg/m2 + cisplatin 20 mg/m2 weekly + radiotherapy 44 Gray (Gy) for 4 weeks).
  4-6 weeks after completion of chemoradiation patients undergo Ivor Lewis esophagogastrectomy.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin; Drug: Fluorouracil; Radiation: chemoradiotherapy; Procedure: Ivor Lewis esophagogastrectomy

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is used in two cycles of neoadjuvant chemotherapy and concomitant chemoradiotherapy
  Other Names: chemotherapy
Drug: Cisplatin — Cisplatin is used in two cycles of neoadjuvant chemotherapy and concomitant chemoradiotherapy
  Other Names: chemotherapy
Drug: Fluorouracil — Fluorouracil is used in two cycles of neoadjuvant chemotherapy
  Other Names: chemotherapy
Radiation: chemoradiotherapy — Distant 3D radiotherapy, single dose 2 Gray (Gy), total dose 44Gy.
  Other Names: chemoradiation
Procedure: Ivor Lewis esophagogastrectomy — Open Ivor Lewis esophagogastrectomy

SUMMARY:
This study is conducted to evaluate efficacy and safety of neoadjuvant chemotherapy followed by preoperative chemoradiotherapy in patients with resectable esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
This study is conducted to evaluate efficacy and safety of neoadjuvant chemotherapy followed by preoperative chemoradiotherapy in patients with resectable esophageal squamous cell carcinoma.

Patients with resectable esophageal squamous cell carcinoma receive 2 cycles of neoadjuvant chemotherapy (paclitaxel 175 mg/м2 iv day 1, cisplatin 75 mg/м2 iv day 1, fluorouracil 750 mg/m2/day continuous infusion, day 1-4 every 3 weeks). Patients who do not progress with distant metastases start preoperative chemoradiotherapy (paclitaxel 50 mg/m2 + cisplatin 20 mg/m2 weekly + radiotherapy 44 Gy for 4 weeks).

4-6 weeks after completion of chemoradiation patients undergo Ivor Lewis esophagogastrectomy irrespectively of objective response.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-75
2. Histologically or cytologically confirmed resectable squamous-cell Tumor (T)1-2 node (N)+, T3N0-3 esophageal cancer. Inclusion of patients with morphologically confirmed and potentially resectable supraclavicular lymphnodes (unilateral, less than 1,5 cm in short axis) is allowed
3. No prior antineoplastic treatment
4. Eastern Cooperative Oncology Group (ECOG) status 0-2
5. Adequate organ function, evidenced by laboratory results with no contraindications to chemotherapy

   * absolute neutrophil count ≥ 1,500 х109/l
   * thrombocytes ≥ 100 х 109/l
   * hemoglobin ≥ 90 mg/l
   * creatinine < 115 µmol/л or creatinine clearance ≥ 55 ml/min
   * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 2.5 x upper limit of normal (ULN)
   * alkaline phosphatase (ALP) > 5 x ULN
   * bilirubin > 1,5 х ULN
6. Women of childbearing potential must have negative pregnancy test, performed 7 days prior to initial treatment
7. Patients must follow appropriate contraception rules during whole treatment period
8. Decrease of body weight must not be more than 20% in last 6 months

Exclusion Criteria:

1. Presence of distant metastases except for metastatic supraclavicular lymphnodes;
2. Bulky (>3 cm) regional lymphnodes metastases;
3. Cervical esophageal cancer;
4. Presence of tumor fistula;
5. Prior malignant tumor, except for proper treated skin basal cell carcinoma and in situ cervical cancer;
6. Active infectious diseases and concomitant diseases that can affect treatment tolerability, surgery and other study procedures;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-07-10 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 24 months
  Disease free survival will be calculated from the start of the treatment to the disease progression or death of any reason.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall survival will be calculated from the start of the treatment to the death of any reason.
Objective response rate according to RECIST 1.1 | 24 months
  Objective response rate will be evaluated separately after chemotherapy and chemoradiotherapy.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 24 months
  Toxicity will be assessed separately after chemotherapy, chemoradiotherapy and surgery according NCI CTC AE 4.0
Pathological complete response rate following chemoradiotherapy | 24 months
  Pathological complete response rate following chemoradiotherapy will be assessed in resected patients

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Tryakin, MD, PhD, Principal Investigator — N.N.Blokhin Russian Cancer Research Center
Locations (2):
- Russia (2):
  - Alexey Tryakin, Moscow
  - Russian Cancer Research Center named after N.N.Blokhin RAMS, Moscow

IPD SHARING:
Plan to Share IPD: Undecided